CLINICAL TRIAL: NCT05168020
Title: Evaluation of a Self-Monitoring Intervention to Reduce Safety Behaviors in Social Anxiety: A Randomized Controlled Trial
Brief Title: Evaluation of a Self-Monitoring Intervention to Reduce Safety Behavior in Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002247
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Social Anxiety
Keywords: Social Anxiety; Safety Behaviors; Intervention; Text-message

STUDY DESIGN:
Intervention Model Description: Participants are randomized in to one of two conditions
Who Masked: Participant
Masking Description: Participants will receive one of two matched interventions. They will not be told whether they are receiving the active or control intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Fading (Experimental): Participants will be asked to identify their five most common SBs from the SAFE. Participants will then be shown a sample checklist with instructions to fill it out. For the next 14 days, participants will receive the following text message "Please remember to avoid using SBs you selected. As you drop them, you'll be able to go into social situations with greater confidence!" with a link for their daily checklist to complete. Participants will be asked to rate how often they engaged in each SB over the past 24 hours
  Interventions: Behavioral: Safety Behavior Fading for Social Anxiety
- Unhealthy Behavior Fading (Active Comparator): Participants will be asked to pick five unhealthy behaviors they engage in most often to decrease. Participants will then be shown the same sample checklist as the Safety Behavior Fading Group. For the next 14 days participants will receive the following text message "Please try to remember to decrease your unhealthy behaviors. As you decrease them you will feel better, and you'll be able to go into social situations with greater confidence!" with a link for their daily checklist to complete. Participants will be asked to rate how often they engaged in each Unhealthy Behavior over the past 24 hours.
  Interventions: Behavioral: Unhealthy Behavior Fading

INTERVENTIONS:
Behavioral: Safety Behavior Fading for Social Anxiety — Participants are asked to reduce or eliminate safety behaviors via text message reminders and checklists to monitor progress
  Arms: Safety Behavior Fading
Behavioral: Unhealthy Behavior Fading — Participants are asked to reduce or eliminate unhealthy behaviors via text message reminders and checklists to monitor progress
  Arms: Unhealthy Behavior Fading

SUMMARY:
The current study aims to explore the efficacy of a text message based Safety Behavior Fading Intervention compared to an active control intervention.

DETAILED DESCRIPTION:
Safety behavior fading may be a viable standalone intervention for social anxiety. In the present trial, participants high in social anxiety will be randomized to either receive a daily checklist exercise aimed at eliminating (1) safety behaviors or (2) unhealthy behaviors. Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their four most habitual social anxiety safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day. Individuals randomly assigned to the control condition will receive similar text messages and a daily checklist to encourage fading of unhealthy behaviors. Participants in both conditions will complete checklists for 28 days. After day 14 of treatment, participants will re-select their target safety behaviors or unhealthy behaviors, and will then be prompted to reduce these new behaviors for another 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Social Phobia Inventory Score >29
* Stable Psychotropic Medications for 4 weeks prior to participation

Exclusion Criteria:

* Currently participating in psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Change in Social Phobia Inventory Score | Day 0, Day 14, Day 42
  Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT05168020/Prot_000.pdf
  • Informed Consent Form (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT05168020/ICF_001.pdf